CLINICAL TRIAL: NCT07365189
Title: Effectiveness of the Online Video-feedback Intervention to Promote Positive Parenting and Sensitive Discipline (Online VIPP-SD). A Randomized Control Trial in Chile
Brief Title: Online Parenting Support With VIPP-SD in Chile
Acronym: VIPP-SD Chile
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad San Sebastián (Other)
Responsible Party: Principal Investigator, RODRIGO ALEJANDRO CARCAMO LEIVA, Full Professor, Universidad San Sebastián
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CEC N°69-25; 1252183 (Other Grant/Funding Number: FONDECYT)
Record Dates: First submitted 2025-11-20; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Parents; Burnout
Keywords: VIPP-SD online; maternal sensitivity; parental burnout; infant attachment; parental limit-setting
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Families in the control group will be contacted online individually by a psychologist (different from interveners) six times to discuss parenting strategies and child development, serving as an active control group. Later, they will receive the online VIPP-SD intervention in the experimental group by the same group of interveners.
- Experimental Group (Experimental): The intervention is delivered through a videoconference platform that allows 1) to record the parent-child tasks and 2) to simultaneously share the previously recorded parent- child interaction and provide feedback. The intervener provides directions in the recording sessions that ensure clearly capturing parent and child facial expressions during the task. Moreover, considering the delivery format, it is essential that both parents and interveners have access to good-quality internet and an electronic device (mobile phone, computer, tablet) with camera. To prevent fatigue arising from the delivery format, it was decided to shorten the sessions, with 30-minute sessions for recording the parent-child task and 40-60-minute sessions for video reviewing and feedback. Thus, Online-VIPP has 12 sessions with alternating recording sessions and video feedback sessions.
  Interventions: Behavioral: Video Intervention to Promote Positive Parenting and sensitive discipline (VIPP-SD)

INTERVENTIONS:
Behavioral: Video Intervention to Promote Positive Parenting and sensitive discipline (VIPP-SD) — The intervention is delivered through a videoconference platform that allows 1) to record the parent-child tasks and 2) to simultaneously share the previously recorded parent- child interaction and provide feedback. The intervener provides directions in the recording sessions that ensure clearly capturing parent and child facial expressions during the task. Moreover, considering the delivery format, it is essential that both parents and interveners have access to good-quality internet and an electronic device (mobile phone, computer, tablet) with camera. To prevent fatigue arising from the delivery format, it was decided to shorten the sessions, with 30-minute sessions for recording the parent-child task and 40-60-minute sessions for video reviewing and feedback. Thus, Online-VIPP has 12 sessions with alternating recording sessions and video feedback sessions.
  Arms: Experimental Group

SUMMARY:
The goal of this randomized controlled trial is to test whether the online Video-feedback Intervention to Promote Positive Parenting and Sensitive Discipline (VIPP-SD) can reduce parental burnout and improve parenting practices, in mothers of young children in Chile.

The main questions it aims to answer are:

* Does the online VIPP-SD increase maternal sensitivity and the use of consistent but gentle limit setting?
* Does it reduce parental burnout?
* Does it improve parental stress and child attachment security and reduce child conduct problems? Researchers will compare families who receive the online VIPP-SD to families in a waitlist control group with dummy treatment to see if VIPP-SD has benefits for parents and children.

Participants will be mothers of children aged 11-16 months at the start of the study who report elevated levels of parental burnout. Mothers in the intervention group will:

* Take part in 12 weekly online sessions with a trained intervener
* Receive video-feedback on their own interactions with their child
* Learn strategies to respond sensitively to their child's needs and to use positive discipline The study will also measure potential moderators such as maternal mental health, child temperament, and family sociodemographic factors.

ELIGIBILITY:
Inclusion Criteria:

* Mothers >18 years
* Child age between 11 - 16 months old at first contact
* Mothers scoring in the top 30% of our sample on the Parental Burnout Scale (BPPS)
* Written informed consent of mothers as participants and guardians
* Internet connection at mother's home.

Exclusion Criteria:

* Child or parent with severe sensory impairment, learning disability, or language limitation
* Sibling already participating in the trial
* Family participating in active family court proceedings
* Parent participating in another closely related research trial and/or receiving an individual video-feedback intervention.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — inclusion criteria:
  * Mothers >18 years
  * Child age between 11 - 16 months old at first contact
Enrollment: 140 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-03-30 (Estimated)

PRIMARY OUTCOMES:
Maternal sensitivity | Pre-test (pre-intervention for the experimental group and at the same time for the control group), and post-test (1 month after the end of the intervention).
  The Ainsworth et al. sensitivity scale will be used to measure maternal sensitivity in a 10-minute free play session. Trained observers code the caregiver's behavior using two rating scales: Sensitivity vs. Insensitivity and Cooperation vs. Intrusiveness, on a scale ranging from 1 to 9, with high values indicating greater sensitivity and cooperation. The procedure will be applied twice, first in the pre-test at home and again in the post-test in the laboratory.
Maternal Limit Setting | Pre-test (pre-intervention for the experimental group and at the same time for the control group), and post-test (1 month after the end of the intervention).
  Parental limit-setting will be observed in a don't touch task. The task is video-taped and parental limit- setting is coded for positive discipline, using an adapted version of the revised Erickson 7-point rating scale for supportive presence, physical interference, rated on a 5-point scale, and Laxness, rated on a 5-point scale.
Parental Burnout | Pre-test (pre-intervention for the experimental group and at the same time for the control group), and posttest (1 month after the end of the intervention).
  The Parental Burnout Assessment (PBA) is a 23-item questionnaire measuring the four dimensions of parental burnout: exhaustion - physical and emotional tiredness, contrast - the perceived discrepancy between the ideal caregiver they would like to be and the one they are currently, a comparison that produces guilt, feelings of being fed up - feeling tired of the parental role, and emotional distancing - putting an affective distance between themselves and their children). The Likert scale response options are: "never" (0), "a few times a year or less" (1), "once a month or less" (2), "a few times a month" (3), "once a week" (4), "a few times a week" (5), "every day" (6). High scores imply high levels of parental burnout.
Fidelity of the Online VIPP-SD | Immediately after the intervention
  Based on written and audio-recorded feedback of sessions, fidelity will be coded in terms of the delivery of key components of the treatment, as well as global adherence to the manual. Note that fidelity is promoted by regular intervision and supervision sessions. We will randomly select 10% of audio recordings for two assessors trained in the intervention to rate the adherence to the VIPP-SD manual using a 5-point scale (1 = Did not follow the manual at all, 2 = Adapted most of the material, did not follow the manual closely, 3 = Sometimes adapted the material, followed manual somewhat, 4 = Adapted only minor elements, followed the manual quite closely, and 5 = Followed the manual very closely and delivered the session as specified). A score of 3 will be set as the acceptable fidelity threshold, as to receive this score most core components of the intervention are present in the feedback.

SECONDARY OUTCOMES:
Hair Cortisol Concentrations | Pre-test (pre-intervention for the experimental group and at the same time for the control group), and post-test (1 month after the end of the intervention).
  Hair samples will be collected by a trained research assistant. As hair grows approximately 1 cm per month (4 cm at least per sample), every 1 cm segment of hair represents the past month. To collect hair samples, a strain of hair at the base of the vertex posterior of the scalp is selected and cut right at the scalp. Hair samples will be put into foil and stored at a dark location at room-temperature until sent to the lab for analysis.
Child Conduct Problems | Pre-test (pre-intervention for the experimental group and at the same time for the control group), and post-test (1 month after the end of the intervention)
  Child conduct problems will be measured using the parent-reported Child Behavior Checklist (CBCL) at the pre- and posttest. The CBCL is a 100-item questionnaire that asks parents to rate how true the behavior is of their child over the last two months on a three-point scale (0 = not true, 1 = somewhat true, or 2 = very true or often true). The measure gives a total score, and scores for externalizing and internalizing behavior problems. The externalizing score is made up of scores for attention problems and aggressive behaviors. We will use the aggresive behaviors subscale to evaluate child conduct problems. This measure will additionally be used in the economic evaluation.
Infant attachment security | Post-test (1 month after the end of the intervention).
  The Strange Situation Procedure (SSP), considered the "gold standard measure" for the assessment of infant attachment pattern in a laboratory procedure, will be used at the post-test. The SSP consists of a series of eight episodes in which the child is exposed to stressful situations such as the entry of a stranger into the room and brief separation from the caregiver, alternating with meetings with the caregiver. The procedure is conducted in a one-way laboratory room set up as a living room with toys and requires recording for later coding. For the attachment outcome, the coding will be based on the continuous scale of security, secure v/s insecure dichotomic classifications, and the D-scale.
Health and social care service use | Pre-test (pre-intervention for the experimental group and at the same time for the control group), and post-test (1 month after the end of the intervention)
  Health and social care service use in experimental and control groups will be measured using the Child and Adolescent Service Use Schedule (CA-SUS). Parents report their own and their child's use of accommodation, hospital, community health and social services, and prescribed medication. This measure will be used for economic evaluation.
Parent's quality of life | Pre-test (pre-intervention for the experimental group and at the same time for the control group), and post-test (1 month after the end of the intervention)
  Quality of life will be measured with the 36-Item Short Form Health Survey questionnaire (SF-36). The SF-36 is a self-report questionnaire assessing health-related quality of life across eight physical and mental health domains. This measure will be used for economic evaluation.

OTHER OUTCOMES:
Parental depression and anxiety symptoms | Pre-test (pre-intervention for the experimental group and at the same time for the control group), and post-test (1 month after the end of the intervention).
  Description: Two subscales of the Brief Symptom Inventory (BSI) will be used to assess depression and anxiety symptoms of both parents. Each subscale has 6 items, which are answered on a 5-point Likert scale according to the frequency of symptomatology within the last seven days, where (0) is Not at all and (4) is Very much.
Temperament | pre-test (pre-intervention for the experimental group and at the same time for the control group).
  The child's temperament will be assessed through the Infant Behavior Questionnaire - Revised - Very Short Form (IBQ-R-VSF) scale in the Spanish version, translated and validated in our country by Farkas & Vallotton, reaching good reliability. The IBQ-R-VSF is a 34-item parent-report questionnaire, which asks about the frequency of occurrence of specific child behaviors during the last week, on a 7-point Likert scale. Scores are obtained on three dimensions: surgency, effortful control and negative affect, where higher scores indicate greater intensity of the dimension.
Parental sleep quality | Pre-test (pre-intervention for the experimental group and at the same time for the control group), and posttest (1 month after the end of the intervention).
  The Pittsburgh Sleep Quality Index (PSQI) will be used to assess parental sleep quality, an important covariate in the burnout literature. The PSQI is a 19-item self-report questionnaire that includes different dimensions of sleep such as sleep disturbances, use of sleep medication, sleep duration and subjective sleep quality. It provides cut-off scores that distinguish between good and poor sleepers.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo A. Cárcamo, Ph.D., Principal Investigator — Facultad de Psicología y Humanidades, Universidad San Sebastián

IPD SHARING:
Plan to Share IPD: Yes
What IPD will be shared: De-identified individual participant data, including primary and secondary outcome measures (maternal sensitivity, parental burnout, physiological stress, child conduct problems, and attachment security), along with key sociodemographic variables. The study protocol and statistical analysis plan will also be shared.
  When: Data will be made available within 12 months after the last publication on the main findings and for up to 5 years following study completion, after reasonable request.
  How: Data will be deposited in an open-access repository (e.g., OSF or institutional repository) or made available upon reasonable request to the principal investigator, subject to approval of a data use agreement ensuring confidentiality and use only for scientific purposes.

REFERENCES:
- [Background] van Ijzendoorn MH, Stevens E, Bakermans-Kranenburg MJ. Development of the virtual-VIPP and a systematic review of online support for families during the COVID-19 pandemic. Attach Hum Dev. 2023 Apr;25(2):223-239. doi: 10.1080/14616734.2023.2179575. PMID 37014109
- [Background] van IJzendoorn MH, Schuengel C, Wang Q, Bakermans-Kranenburg MJ. Improving parenting, child attachment, and externalizing behaviors: Meta-analysis of the first 25 randomized controlled trials on the effects of Video-feedback Intervention to promote Positive Parenting and Sensitive Discipline. Dev Psychopathol. 2023 Feb;35(1):241-256. doi: 10.1017/S0954579421001462. Epub 2022 Jan 17. PMID 35034668